CLINICAL TRIAL: NCT06501573
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Single Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered SGB-9768 in Healthy Volunteers
Brief Title: A Study of SGB-9768 in Adult Healthy Volunteers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Sanegene Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-9768-002
Record Dates: First submitted 2024-07-09; First posted 2024-07-15 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-07

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SGB-9768 (Experimental): a single dose of SGB-9768 by subcutaneous (sc) injection
  Interventions: Drug: SGB-9768
- Placebo (Placebo Comparator): placebo calculated volume to match active treatment by sc injection
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: SGB-9768 — SGB-9768 for sc injection
  Arms: SGB-9768
Other: Placebo — sterile normal saline (0.9% NaCl) for sc injection
  Arms: Placebo

SUMMARY:
This study is a randomized, double-blind, placebo-controlled single ascending dose study of SGB-9768 in healthy volunteers. The purpose is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of subcutaneously administered SGB-9768.

DETAILED DESCRIPTION:
It is a phase 1, randomized, double-blind, placebo-controlled single ascending dose study of SGB-9768. The primary objective is to evaluate the safety, tolerability of SGB-9768 when administered subcutaneously as a single dose to healthy volunteers. The secondary objective is to characterize the pharmacokinetics and pharmacodynamics of subcutaneously administered SGB-9768 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects aged 18 to 55 years are included at the time of informed consent.
* Body mass index between 18 and 28 kg/m2 at screening, inclusive, at screening a weight of at least 45 kg for female and 50 kg for male.
* Physical examination, vital signs, 12-lead electrocardiogram, and laboratory tests be normal or slightly abnormal but not clinically significant according to investigator's judgement.
* Women of child-bearing potential who are not exclusively in same-sex relationships and males with partners of child-bearing potential must agree to use adequate contraception from signing the informed consent until 12 weeks after completion of the follow-up visit.
* Willing to comply with the protocol required visit schedule and visit requirements and provide written informed consent.

Exclusion Criteria:

* A history of or current surgical or medical condition that, in the opinion of the Investigator, may put the subject at significant risk (according to Investigator's judgment) or interfere with the subject's participation in the clinical study.
* History of or evidence of tuberculosis.
* History of recurrent or chronic infections.
* Subjects with a history of meningococcal infection, or subjects who are exposed to Neisseria meningitidis.
* History of asplenia or splenectomy.
* History of abnormalities in complement or hereditary complement deficiency.
* Received an investigational agent within 30 days or 5-half-lives (whichever is longer) before the first dose of the study drug or being in other clinical study.
* History or clinical evidence of drug abuse within 12 months before screening or positive screen for drugs of abuse.
* Used prescribed or over-the-counter medication within 14 days or 5 half-lives (whichever is longer) before the first dose of the study drug unless determined not clinically relevant by the Investigator.
* Any conditions which, in the opinion of the Investigator, would make the subject unsuitable for enrollment or could interfere with the subject's participation in or completion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-05-03 (Estimated); Study Completion 2025-10-17 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of SGB-9768 | 169 days
  Number of Participants with Adverse Events (AEs) and/or Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Pharmacokinetics-Cmax | 48 hours
  Maximum Observed Plasma Concentration (Cmax)
Pharmacokinetics-Tmax | 48 hours
  Time at which the maximum plasma concentration (Cmax) occurs
Pharmacokinetics-AUClast | 48 hours
  Area under the plasma concentration-time curve from dosing (time zero) to the time of the last measured concentration
Pharmacokinetics-AUCinf | 48 hours
  Area Under the Plasma Concentration Versus Time Curve from Zero Extrapolated to Infinity (AUCinf)
Pharmacokinetics-t1/2 | 48 hours
  Terminal Elimination Half-Life (t1/2)
Pharmacokinetics-CL/F | 48 hours
  Total Body Clearance
Pharmacokinetics-Vz/F | 48 hours
  Volume of Distribution (Vz/F)
Pharmacodynamics-C3 | 169 days
  Change From Baseline in Complement 3 (C3)
Pharmacodynamics-complement acitvity | 169 days
  Change From Baseline in Complement Activity

CONTACTS AND LOCATIONS:
Locations (1):
- Huashan hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No